CLINICAL TRIAL: NCT04741360
Title: Improving New Learning and Memory in School Aged Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: New Jersey Commission on Brain Injury Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-987-17
Record Dates: First submitted 2021-02-03; First posted 2021-02-05 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Traumatic Brain Injury
Keywords: Pediatrics
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Story Memory Technique (Experimental)
  Interventions: Other: Modified Story Memory Technique
- Control (Other)
  Interventions: Other: Modified Story Memory Technique

INTERVENTIONS:
Other: Modified Story Memory Technique — 10-session computerized program to improve new learning and memory

SUMMARY:
The currently proposed study addresses a critical need in the clinical care of school-aged children with TBI through the modification of an existing, proven efficacious treatment protocol for learning and memory deficits in persons with moderate to severe TBI, the modified Story Memory Technique (mSMT), as well as the conduct of a pilot double blind, placebo-controlled, RCT of this new pediatric adaptation of the mSMT. Over a decade of research and development conducted at our center has demonstrated the mSMT to be effective for improving new learning and memory in adults with TBI, across three realms of functioning: objective behavior, brain functioning and everyday life. This convincing data provides Class I evidence supporting the efficacy of the mSMT for improving new learning and memory in adults with TBI. Clinical applications around the world have equally attested to its utility in the clinical care of adults with TBI. This highlights the tremendous potential of the mSMT to vastly improve the everyday lives and educational successes of children and adoles-cents living with TBI and the resultant learning and memory deficits. The currently proposed pilot work will begin to document that efficacy. The results of this study therefore have the potential to change clinical practice, inform policy, and improve the lives of children and adolescents living with TBI.

DETAILED DESCRIPTION:
The currently proposed study addresses a critical need in the clinical care of school-aged children with TBI through the modification of an existing, proven efficacious treatment protocol for learning and memory deficits in persons with moderate to severe TBI, the modified Story Memory Technique (mSMT), as well as the conduct of a pilot double blind, placebo-controlled, RCT of this new pediatric adaptation of the mSMT. Over a decade of research and development conducted at our center has demonstrated the mSMT to be effective for improving new learning and memory in adults with TBI, across three realms of functioning: objective behavior, brain functioning and everyday life. This convincing data provides Class I evidence supporting the efficacy of the mSMT for improving new learning and memory in adults with TBI. Clinical applications around the world have equally attested to its utility in the clinical care of adults with TBI. This highlights the tremendous potential of the mSMT to vastly improve the everyday lives and educational successes of children and adoles-cents living with TBI and the resultant learning and memory deficits. The currently proposed pilot work will begin to document that efficacy. The results of this study therefore have the potential to change clinical practice, inform policy, and improve the lives of children and adolescents living with TBI.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 9 and 17.
* Have sustained a TBI at least 1 year ago, that has affected his or her memory.
* Be able to speak and read English fluently.

Exclusion Criteria:

* Diagnosis of MS, or neurological injury or disease in the past (like brain tumor or epilepsy).
* History of significant psychiatric illness (like bipolar disorder, schizophrenia or psychosis).
* Uncontrolled seizures or other unstable medical complications.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
CVLT-C Learning Slope | 6 months
  Memory

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No